CLINICAL TRIAL: NCT03264196
Title: Condylar Head Operative or Conservative 1, Randomised Controlled Trial
Brief Title: Condylar Head Operative or Conservative 1
Acronym: CHOC1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Niall Mcleod, Consultant Oral and Maxillofacial Surgeon, Oxford University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12513
Record Dates: First submitted 2017-08-21; First posted 2017-08-29 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Condylar Process of Mandible Open Fracture
Keywords: condylar hear; fracture; randomised controlled trial
MeSH Terms: conditions — Fractures, Bone | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operative (Active Comparator): Open Reduction and Internal Fixation of Condylar Head Fracture
  Interventions: Procedure: Open Reduction and Internal Fixation
- Conservative (No Intervention): Non-operatively managed Condylar Head Fracture

INTERVENTIONS:
Procedure: Open Reduction and Internal Fixation — Surgical treatment of fracture
  Arms: Operative

SUMMARY:
The condylar head is the part of the lower jaw which forms the joint. Displaced fractures of this area are uncommon but can cause problems with function, such as chewing, if not treated effectively. The medical literature does not have a clear consensus on whether these should be treated operatively (with surgery to reduce and fix the fracture) or conservatively (with advice and exercise and no surgery). The investigators propose a randomised controlled trial comparing the outcome of the operative or conservative treatment of condylar head fractures of the mandible, primarily with regards to patient related outcome measures of mandibular function, and secondarily objective measures of mandibular movement, function and symptoms to try and provide a clearer answer as to the best way of managing them.

DETAILED DESCRIPTION:
The current medical literature provides conflicting evidence as to the benefits of operative or conservative management of displaced condylar head fractures. Whilst conservative treatment has few risks in itself, most of the evidence would suggest that outcomes are not quite as good as operative management. Operative treatment has complications that are not presented by conservative treatment, such as the risk of infection or facial nerve injury and therefore it is important to demonstrate that such treatment has sufficient benefits to merit it's consideration, and to properly inform the patients about the benefits and risks of treatment. When patients present with these injuries it is currently difficult to provide them with good evidence for them to make an informed decision with, as to whether to undergo surgery or not. At present the patient is expected to make a decision as to whether to have surgery or not based on this limited knowledge, and it is the investigator's experience with consulting these patients and the questions they asked that has demonstrated the need for and guided the design of the trial focusing on a patient related outcome quality of life measure, rather than the common objective measures.#

The main purpose of undertaking this RCT is to directly compare the results of operative and conservative management focusing on an outcome which is determined by the patients perception of their function and quality of life rather than purely objective measurements. A randomised controlled trial would provide the strongest level of evidence to support future care decisions and any patient with a unilateral fracture would be considered for inclusion if they can give informed consent and are able to complete the PROM questionnaire at the necessary time points. Exclusion criteria are limited, but include bilateral fractures because these are less common and the results may not be directly comparable.

The trial design has been kept simple and adds no significant burden to patients as all aspects of care and follow up are the same as the current standard of care apart from the completion of the questionnaire, which can be completed relatively quickly during participant's clinic appointments. The investigators are experienced surgeons in this field and able to fully answer any questions from patients with regards to the trial, and to risks and benefits of either treatment option. Neither has any conflict of interest in undertaking the trial.

All trial data will be handled confidentially in line with good governance procedures, and will be monitored by appropriate persons from the trial sponsors.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* Male or Female, aged 18 years or above.
* Be in good health - suitable for general anaesthesia for surgical treatment
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the trial.
* Unilateral condylar head fracture with or without other mandibular body or angle fractures, or other maxillofacial injuries
* Condylar head fracture displaced by at least 2 mm measured on coronal or sagittal CT scan
* In the Investigator's opinion, is able and willing to comply with all trial requirements.

Exclusion Criteria:

* Undisplaced condylar head fractures, or displaced less than 2 mm on coronal or sagittal CT
* Bilateral condylar head fractures
* Pre-existing congenital or acquired pathology of the ipsilateral or contralateral temporomandibular joint - including but not limited to ankylosis, inflammatory arthropathy, idiopathic condylar resorption
* Pregnancy (increased risk of joint pain and laxity)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Difference in functional self reported outcome measure | 12 months
  Difference in function assessed using Mandibular Functional Impairment Questionnaire

SECONDARY OUTCOMES:
Fracture Reduction | 12 months
  Post operative fracture reduction (ramus / condyle height - fracture side compared to normal on post operative OPG)
Mouth Opening | 12 months
  Mean interincisal opening- mm
Mandibular lateral movements | 12 months
  Mean lateral excursion from affected side - mm
Mandibular protrusion | 12 months
  Mean Protrusion - mm
Pain Score | 12 months
  Pain - linkart score (0-10)
Dietary interference | 12 months
  Dietary interference - linkart score (0-10)
Mandibular functional impairment | 12 months
  Functional impairment rating scale (1-4)

CONTACTS AND LOCATIONS:
Overall Officials: Niall MH Mcleod, FRCS(OMFS), Principal Investigator — Oxford University Hospitals
Locations (2):
- United Kingdom (2):
  - University Hospital Coventry, Coventry, Warwickshire
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No